CLINICAL TRIAL: NCT06963086
Title: Implementing an Eating Disorder Prevention Program for Youth in Nova Scotia
Acronym: EDPP-P2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Susan Gamberg (Other)
Collaborators: Queen Elizabeth II Health Sciences Centre Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Susan Gamberg, Registered psychologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EDPP-P2
Record Dates: First submitted 2025-04-21; First posted 2025-05-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Body Image; Body Dissatisfaction; Dietary Restraint; Negative Affect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the Body Project (Experimental)
  Interventions: Behavioral: Eating disorder prevention program (the Body Project)

INTERVENTIONS:
Behavioral: Eating disorder prevention program (the Body Project) — The Body Project is an eating disorder prevention program for girls and young women aged 15-22 years old. The program will be delivered in groups of 6-10 youth by peer mentors, and in two formats: in-person and virtual. We are assessing two versions of the program - a 6-session version (6 weekly 45-minute sessions) and a 2-session version (2 weekly 2-hour sessions). Participants will be divided into 4 cohorts: high school in-person, university in-person, high school-aged (15-18 years) virtual, and university-aged (19-22 years) virtual. The high school in-person groups will do the 6-session version, and the university in-person groups as well as all virtual groups will do 2 weekly 2-hour sessions. Both versions cover similar content, and use a scripted intervention manual.

SUMMARY:
The goal of this study is to evaluate the Body Project, which is an eating disorder prevention program for youth 15-22 years old. The main question it aims to answer is 'Can an eating disorder prevention program, specifically the Body Project, be successfully delivered to youth in Nova Scotia'?

This study will determine the feasibility of implementing the Body Project in Nova Scotia by assessing the following objectives:

1. Acceptability (how well the Body Project is received by, and the extent to which it is perceived as meeting the needs of, youth in Nova Scotia).
2. Demand (the extent to which youth in Nova Scotia are interested in and willing to engage with the program).
3. Integration (the extent to which the Body Project is judged as feasible by the group facilitators).
4. Effectiveness (the extent to which the Body Project reduces eating disorder risk factors in youth in Nova Scotia).

Participants will:

* Attend a total of 4-4.5 hours of Body Project group sessions, which are led by peer mentors.
* Complete outcome measure questionnaires before their first session and after their last session.
* Participate in a focus group with their session group members after their last session.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a girl/woman.
* Be between the ages of 15-22 years old.
* For inclusion in an in-person group, an individual must be currently enrolled as a student at the school where they will participate in sessions.
* For inclusion in a virtual BP group, an individual must live in and/or attend school in Nova Scotia, and have access to a computer (e.g., laptop, desktop computer, cellphone) with internet connection and a webcam that can be used in a private location (if a participant does not have a private location to use when attending sessions, they will be asked to wear headphones).
* Able to complete English computer-based self-report questionnaires (with adequate accommodation, if necessary).
* Provides informed consent (or verbal assent with informed consent provided by parent/guardian).

Exclusion Criteria:

* Previous participation in the Body Project.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Eligible individuals are those who self-identify as a girl or woman.
Enrollment: 120 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the Body Project as measured with focus groups | Immediately following completion of the final Body Project session for each group (week 2 for university and virtual groups; or week 6 for high school in-person groups)
  All participants will complete a focus group with their fellow Body Project group members immediately following their final session. The focus group will follow a semi-structured guide based on a framework for assessing acceptability of health interventions.

SECONDARY OUTCOMES:
Acceptability of the Body Project as measured with program dropout rate | From a participant's first session (week 1) to last session (either week 2 or week 6, depending on group).
  Participants will be coded as a 'dropout' from the intervention if they stop attending sessions (determined with session attendance records from group facilitators). Acceptability based on dropout rate will be indicated if the dropout rate in the final session is equal to, or less than, the 20-30% rate reported in effectiveness trials for the BP.
Acceptability of the Body Project as measured with a questionnaire on participant satisfaction with the program | After a participant's last session (either week 2 or week 6, depending on group).
  Acceptability in terms of satisfaction with the program will be measured using an investigator-created questionnaire based on the Client Satisfaction Questionnaire - an 8-item self-report measure of the quality and effectiveness of a health service. Item responses are on a 4-point scale. Scores range from 8-32, with higher scores indicating higher satisfaction. Acceptability based on satisfaction questionnaire scores will be demonstrated if participants, on average, report at least moderate satisfaction (defined as a score of 24).
Demand for the Body Project as measured with recruitment rate | At 24 months after recruitment begins.
  Demand feasibility will be met if there are enough participants to run 3-5 rounds of Body Project groups per cohort (totaling 96-120 youth) during the recruitment period.
Effectiveness of the Body Project for reducing pursuit of the thin ideal as measured with the Thin-Ideal Internalization Scale (TIIS) | From baseline to after a participant's last session (either week 2 or week 6, depending on group).
  The TIIS is the modernized version of the Ideal Body Stereotype Scale and is an 8-item self-report measure assessing internalization of the thin beauty ideal. Response options range from 1 = strongly disagree to 5 = strongly agree. Scores range from 8-40, with higher scores indicating higher internalization of the thin ideal. Feasibility will be met if there are significant within-group reductions of at least a moderate effect size (Cohen's d > 0.5).
Effectiveness of the Body Project for reducing body dissatisfaction as measured with the Satisfaction and Dissatisfaction with Body Parts Scale (SDBPS) | From baseline to after a participant's last session (either week 2 or week 6, depending on group).
  Nine items from the Body Image Satisfaction Scale will be used to assess satisfaction with nine body parts, in line with previous Body Project research. Responses range from 1 = extremely satisfied to 6 = extremely dissatisfied. Scores range from 9-54, with higher scores indicating greater dissatisfaction. Feasibility will be met if there are significant within-group reductions of at least a moderate effect size (Cohen's d > 0.5).
Effectiveness of the Body Project for reducing negative affect as measured with the Positive Affect and Negative Affect Scale-Revised (PANAS-X) | From baseline to after a participant's last session (either week 2 or week 6, depending on group).
  In line with previous BP research, 20 items from the PANAS-X subscales for sadness, guilt, and fear/anxiety will be used to assess negative affect. Responses range from 1 = not at all to 5 = extremely. Scores range from 20-100, with higher scores indicating greater negative affect. Feasibility will be met if there are significant within-group reductions of at least a moderate effect size (Cohen's d > 0.5).
Effectiveness of the Body Project for reducing disordered eating behaviors and attitudes as measured with the Eating Disorder Examination Questionnaire (EDE-Q) | From baseline to after a participant's last session (either week 2 or week 6, depending on group).
  The EDE-Q global score is calculated from 22 attitudinal questions regarding eating restraint and concerns, weight concerns, and shape concerns. EDE-Q global scores range from 0-6, with higher scores indicating increased severity of ED psychopathology. Feasibility will be met if there are significant within-group reductions of at least a moderate effect size (Cohen's d > 0.5).

OTHER OUTCOMES:
Integration of the Body Project as assessed with group facilitator surveys | After a facilitator has completed their last session (at study completion - about 24 months after recruitment starts).
  Facilitators will complete an open-ended feedback survey to ascertain what went well, what alterations (if any) are needed, and what barriers facilitators encountered or identified.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Gamberg, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Abbie J Lane Memorial Building, QEII Health Sciences Centre, Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963